CLINICAL TRIAL: NCT05149365
Title: Sitagliptin Efficacy and Safety for Prevention of Acute Graft Versus Host Disease in Patients Receiving Alternative Donor Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Sitagliptin for Prevention of aGVHD After Alternative Donor Transplation
Acronym: SHIELD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); The Second People's Hospital of Huai'an (Other); The First People's Hospital of Changzhou (Other); Xinqiao Hospital of Chongqing (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SZ-GVHD 06
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Acute-graft-versus-host Disease; Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Sitagliptin; Alternative Donor
MeSH Terms: interventions — Sitagliptin Phosphate; Cyclosporine

STUDY DESIGN:
Intervention Model Description: Prospective, Multi-center, Open-label, Randomized, Controlled Clinical Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin Group (Experimental): 95 adult patients with hematologic malignancies receiving Alternative Donor HSCT, who will receive Sitagliptin combined with Standard prophylaxis regimen for GVHD of Alternative Donor HSCT.
  Interventions: Drug: Sitagliptin + Standard Prophylaxis
- Standard Group (Active Comparator): 95 adult patients with hematologic malignancies receiving Alternative Donor HSCT, who will only receive Standard prophylaxis regimen for GVHD of Alternative Donor HSCT
  Interventions: Drug: Standard Prophylaxis

INTERVENTIONS:
Drug: Sitagliptin + Standard Prophylaxis — Sitagliptin 600 mg ever 12 hours orally will be given starting from the day before transplantation through day +14 after transplantation and Standard prophylaxis regimen
  Other Names: Cyclosporine (CsA),Methotrexate (MTX), Mycopherol ester (MMF) and Antithymic Globulin
  Arms: Sitagliptin Group
Drug: Standard Prophylaxis — Standard prophylaxis regimen for GVHD of Alternative Donor HSCT, include Cyclosporine (CsA),Methotrexate (MTX), Mycopherol ester (MMF) and Antithymic Globulin
  Other Names: Cyclosporine (CsA),Methotrexate (MTX), Mycopherol ester (MMF) and Antithymic Globulin
  Arms: Standard Group

SUMMARY:
Primary Objective:

It is hypothesized that the efficacy of Sitagliptin would reduce the incidence of grade II-IV acute Graft Versus Host Disease (GVHD) by day +100 post-transplant in patients undergoing alternative donor (related haploid or unrelated donor ) allogeneic Hematopoietic Stem Cell Transplantation (HSCT) and receiving standard GVHD prophylaxis.

Secondary Objectives

The following descriptive secondary objectives will be studied:

1. Determine the tolerability and potential toxicity of sitagliptin in patients undergoing allogeneic HSCT.
2. Determine the cumulative incidence of grades II-IV acute GVHD by day +100.
3. To investigate the cumulative incidence of grades III-IV acute GVHD.
4. To investigate the engraftment kinetics of absolute neutrophil count and platelets.
5. To evaluate the incidence of Cytomegalovirus (CMV), Epstein-Barr virus (EBV) and other infections occurring during the 100 days post-transplant.
6. To study non-relapse mortality (NRM) at day +100, and 1 year post-transplant.
7. Determine the overall survival at 1 year post-transplant.
8. Determine the incidence of chronic GVHD.
9. Determine the cumulative incidence of relapse of the primary hematological malignancy.

DETAILED DESCRIPTION:
This is a Prospective, Multi-center, Open-label, Randomized, Controlled clinical trial of Sitagliptin for the prevention and safety of aGVHD after Alternative Donor hematopoietic stem cell transplantation.

190 adult patients with hematologic malignancies receiving haploid or unrelated donor sourced HSCT are planned to be enrolled competitively in this study from 5 clinical centers in China. These patients will be randomly assigned to two groups of 95 patients each, which one is experimental group and the other is control group. 95 patients in experimental group will receive Sitagliptin combined with Standard prophylaxis for GVHD. 95 patients in the control group will receive Standard prophylaxis regimen for GVHD of Alternative Donor HSCT.

Control group uses antithymocyte immunoglobulin (ATG)+cyclosporin A (CSA)+MMF+MTX for GVHD prophylaxis with the details as follows: CSA 3mg/kg continuous i.v. drip, start before Day -7, change to p.o. when gastrointestinal function recovers with a dose of 5mg/kg as two divided doses, maintaining CSA within 150-250ng/ml（If CsA cannot be tolerated, tacrolimus may be used as an alternative.）; MTX 15mg/m2,Day +1, 10mg/m2,Days +3, +6, and +11; MMF 0.5g bid, starting from Day -7 to day +30 for one month; ATG 2.5mg/kg/d, Day -4 to Day -1.

Experimental group will take Sitagliptin orally from d-1 to d+14 in addition to Standard Prophylaxis Regimen.

With regard to the content of dose reduction of CSA (including time and reduction rate), it is recommended for patients with hematologic malignancies in standard risk group to start to reduce dose after 3-6 months in the absence of GVHD and reoccurrence. The specific reduction rate can be determined at each site; the patients with GVHD will be managed by routine practice in this site.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 18 to ≤ 60 years
2. Eastern Cooperative Oncology Group (ECOG）score 0-2 points / Karnofsky score ≧80
3. To receive allogeneic hematopoietic stem cell transplantation from related haploid or unrelated donor
4. The pretreatment of modified Bu/Cy+ATG scheme was planned.
5. Patients with malignant hematological diseases indicated by transplantation and in complete remission (CR) state.
6. Expected survival ≥ 3 months
7. Signed written informed consent (Patient must be capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent)
8. Agree to use effective contraception

Exclusion Criteria:

1. Prior allogeneic hematopoietic stem cell transplant
2. Allergy/intolerance to Sitagliptin
3. There are contraindications for Sitagliptin use.
4. Moderate or severe renal insufficiency
5. Patients with diabetes mellitus requiring insulin secretagogues and/or insulin
6. Human immunodeficiency virus or active hepatitis C virus or active hepatitis B virus infection
7. Active infection that is difficult to control
8. Vital organ function cannot tolerate transplantation
9. Other malignant tumors outside the blood system, except the following diseases: malignant tumors that have been cured for 3 years without active lesions; Adequate treatment of non-melanoma skin cancer without active foci of malignant amygdala and carcinoma in situ
10. There is evidence that may interfere with the study or make patients at risk of serious complications or medical conditions, including but not limited to serious cardiovascular diseases (such as New York heart association class III or IV heart disease over the past six months of myocardial infarction, unstable type of cardiac arrhythmias) or unstable angina and/or severe lung disease (e.g. History of severe obstructive pulmonary disease and symptomatic bronchospasm)
11. Pregnant or lactating women
12. Any life-threatening medical condition or organ system dysfunction considered by the investigator may endanger the patient's safety by interfering with the absorption or metabolism of sitagliptin or putting study results at unnecessary risk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Development Grade II-IV Acute GVHD by Day +100 Following Transplantation | up to 100 days
  Percent of patients and the 95% Confidence interval who have Grade II-IV Acute GVHD by 100 days following transplantation. Only patients who were on the study for at least 100 days post transplantation were included in the analysis.

SECONDARY OUTCOMES:
Development Grade II-IV Acute GVHD at Day +100 | 100 days from transplant
  Fine-Gray and Cause-specific COX methods will be used to conduct a competing risk analysis. Time until grade II-IV acute GVHD will be calculated from transplant through grade II-IV acute GVHD or death from GVHD. Patients who relapsed or died from causes other than GVHD will be considered a competing risk population and calculated from time of transplant until relapse or death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage of grade II-IV acute GVHD at day +100 was calculated along with a 95% confidence interval.
Percentage of Patients With Grade III-IV Acute GVHD at Day +100 | 100 days from transplant
  Fine-Gray and Cause-specific COX methods will be used to conduct a competing risk analysis. Time until grade III-IV acute GVHD will be calculated from transplant until grade III-IV acute GVHD or death from GVHD. Patients who relapsed or died from causes other than GVHD will be considered a competing risk and calculated from time of transplant until relapse or death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage of grade II-IV acute GVHD at day +100 was calculated along with a 95% confidence interval.
Cumulative incidence of early transplant-related death (TRM) within 100 days after transplantation | 100 days from transplant
  Percent of patients and the 95% Confidence interval who died within 100 days after transplantation.
Median Time to Engraftment of Neutrophils | up to 1 month
  Time to neutrophil engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of neutrophils is defined as the time from day 0 to the date of the first of three consecutive days after transplantation during which the absolute neutrophils count (ANC) is at least 0.5 x109/l. Patients who did not have neutrophil engraftment before death will be censored at the date of death. The median and 95% confidence intervals were calculated.
Median Time to Engraftment of Platelets | up to 4 months
  Time to platelet engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of platelets is defined as the time from day 0 to the first of seven consecutive Complete Blood Counts (CBCs) obtained on different days after transplantation during which the platelet count is at least 20 x109/l. The CBCs obtained should be at least seven days after the most recent platelet transfusion. The median and 95% confidence intervals were calculated.
Number of Unique Patients With Infections by Day +100 | 100 days from transplant
  Number of unique patients who had each type of infection (i.e., viral, bacterial, fungal, etc.) during the 100 days post transplant. A patient could have more than one type of infection.
Percentage of Patients With Non-relapse Mortality (NRM) at +1 Year | 1 year from transplant
  Kaplan-Meier methods will be used to conduct a competing risk analysis. Time until non-relapse death will be calculated from transplant until death. Patients who died from relapse will be considered a competing risk and calculated from time of transplant until death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage of non-relapse mortality at day +365 was calculated along with a 95% confidence interval.
Percentage of Patients Surviving at +1 Year | 1 year from transplant
  Duration of time from the start of treatment to time of death due to any causes. Patients who do not die will be censored on their last known alive date. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated. The cumulative incidence percentage of survival at day +365 was calculated along with a 95% confidence interval.
Percentage of Patients Diagnosed With Chronic GVHD at 1 Year | 1 year from transplant
  Patients surviving at least 100 days will be evaluable for chronic GVHD. The cumulative incidence of chronic GVHD (total, and mild, moderate, severe) will be described using deaths from causes other than chronic GVHD considered as a competing risk. Kaplan-Meier methods will be used to conduct a competing risk analysis. Time until chronic GVHD will be calculated from transplant until chronic GVHD or death from GVHD. Patients who relapsed or died from causes other than GVHD will be considered a competing risk and calculated from time of transplant until relapse or death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage at 1 year will calculated along with a 95% confidence interval.
Percentage of Patients With Relapse of the Primary Hematological Malignancy at 1 Year | 1 year from transplant
  Kaplan-Meier methods will be used to conduct a competing risk analysis. Time until relapse will be calculated from transplant until relapse or death from relapse. Patients who died from causes other than relapse will be considered a competing risk and calculated from time of transplant until death. Otherwise, patients will be censored and calculated from transplant until the last known alive date. The cumulative incidence percentage of relapse at day +365 was calculated along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, Professor, Principal Investigator — The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China